CLINICAL TRIAL: NCT02097173
Title: Relative Bioavailability of Methotrexate (MTX) 50 mg/mL Administered Subcutaneously (SC) by a Disposable Autoinjector (Metoject® Prefilled Pen) Compared With Intramuscular (IM) Administration of the United States Reference Listed Drug Methotrexate Injection (USP 25 mg/mL [Hospira]) in Patients With Psoriasis
Brief Title: Bioavailability in Patient With Psoriasis: Metoject Prefilled Pen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: medac GmbH (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MC-MTX.12/PK
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SC MTX followed by IM MTX (Other): 1 subcutaneous injection of 30 mg methotrexate administered by a prefilled pen (50mg/mL) followed by 1 intramuscular injection of 30 mg methotrexate (comparator) after a wash-out phase of 1 week
  Interventions: Drug: Methotrexate
- IM MTX followed by SC MTX (Other): 1 intramuscular injection of 30 mg methotrexate (comparator) followed by 1 subcutaneous injection of 30 mg methotrexate by a prefilled pen (50mg/mL) after a wash-out phase of 1 week
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate

SUMMARY:
This study is conducted to assess the relative bioavailability of MTX administered subcutaneously via a prefilled pen (50mg/mL) compared with MTX administered via IM injection (25mg/mL).

ELIGIBILITY:
Inclusion Criteria:

* Is able to understand and follow instructions during the study
* Has a diagnosis of moderate to severe psoriasis based on a dermatologic evaluation
* Provides written informed consent
* Is male or female and is aged 18 to 65 years, inclusive
* Has a body mass index (BMI) within the range 18 through 30 kg/m2.

Main Exclusion Criteria:

* Is receiving concomitant treatment for psoriasis with a biologic or conventional systemic treatments (eg, cyclosporine, azathioprine, fumaric acid esters, Leflunomide), other than MTX every week
* Has used antibiotics within 14 days prior to Screening or requires use prior to study completion
* Has used any of the following medications within 14 days prior to Screening or requires use prior to study completion, unless on a stable, daily dose: Non steroidal antiinflammatory drugs (NSAIDs), Diuretics, Folic Acid, Hydrochloroquine, Probenicid, Proton-pump inhibitors
* Has, other than psoriasis, any uncontrolled cardiac disease, liver disease, lung disease, hematologic disease, gastrointestinal disease, or other systemic disease, that in the opinion of the investigator, would present an unacceptable risk if he or she were to participate in the study
* Has ongoing acute or chronic infection within 14 days prior to Screening
* Has renal insufficiency , hepatic insufficiency, impaired hematopoiesis, known severe, acute, or chronic infection, history of malignancy, history of or suspected abuse of drugs or alcohol
* allergic reactions or serious adverse reactions to the study drug
* Is a female subject who is pregnant, trying to become pregnant, or breast feeding, or of childbearing potential, sexually active and not practicing a highly reliable method of birth control
* Is a male subject with a female partner of childbearing potential, not had a vasectomy and not using a condom and/or cervical cap/diaphragm with spermicide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To determine the relative bioavailability of MTX based on the parent compound MTX when administered by SC injection with a prefilled pen (50 mg/mL) as compared with IM administration (25 mg/mL) | 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials of Texas, Inc., San Antonio, Texas, United States